CLINICAL TRIAL: NCT00503386
Title: A Phase II,Multicenter,Randomized,Double-blind,Cross-over Study of Palonosetron Compared With Granisetron in Prevention of Chemotherapy-induced Nausea and Vomiting in Asian Population
Brief Title: Safety and Efficacy of Palonosetron in Preventing Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Jiuyuan Gene Engineering Co. Ltd., (Industry)
Collaborators: Sun Yat-sen University (Other); Tigermed Consulting Co., Ltd (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HJGene_SYat-sen_06_01
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Nausea; Vomiting; Chemotherapy
Keywords: chemotherapy-induced nausea and vomiting; acute; delayed; emesis; antiemetics; 5-HT3 receptor antagonist; granisetron; palonosetron
MeSH Terms: conditions — Nausea; Vomiting | interventions — Palonosetron; Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Palonosetron
Drug: Granisetron

SUMMARY:
The purpose of this study is to determine whether palonosetron is tolerate and effective in preventing chemotherapy-induced nausea and vomiting in oriental population. The study is comparing the safety and efficacy of palonosetron with granisetron, a frequently used antiemetic in China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 yrs and <70 yrs with histologically or cytologically confirmed
* Malignant disease
* Naive or nonnaive to chemotherapy, with a Karnofsky score of ≥ 60
* Scheduled to receive two courses of moderately emetogenic chemotherapy or cisplatin 60 ~ 80 mg/m2 on study Day 1
* Use of reliable contraceptive measures (for females of childbearing potential) and negative pregnancy test at baseline visit
* Patients with hepatic, renal, or cardiovascular impairment eligible at the investigator's discretion
* Patients experiencing, at maximum, mild nausea after previous chemotherapy eligible at the investigator's discretion
* Predicted life expectancy of ≥ 3 months
* Provision of written informed consent.

Exclusion Criteria:

* Inability to understand or cooperate with study procedures
* Receipt of investigational drugs ≤ 30 days before study entry
* Receipt of other investigational drugs during the course of this study
* Seizure disorder or any condition requiring anticonvulsants, sedatives
* CNS malignancy or metastasis
* Ongoing emesis due to obstruction of digestive tract
* Emesis, retching, or Grade 2 or 3 nausea 24 hrs before chemotherapy
* Moderate or severe nausea and vomiting after any previous chemotherapy
* Scheduled receipt of any chemotherapeutic agent with an emetogenicity level >3 during study Days 2-5
* Scheduled receipt of radiotherapy of the upper abdomen or cranium on study Days 2-5
* Scheduled to receive any other drug with potential antiemetic efficacy within 24 h of study initiation and throughout day 5
* Contraindications to 5-HT3 receptor antagonists
* Contraindications to chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Complete Protection from Vomiting (ie.Complete Response in Preventing Vomiting) | 0-24h, 24-120h , 0-120h following chemotherapy

SECONDARY OUTCOMES:
Major Protection from vomiting | 0-24h,24-120h,0-120h following chemotherapy
Major Protection from nausea | 0-24h,24-120h,0-120h following chemotherapy
Complete Protection from Both Vomiting and Nausea | 0-24h,24-120h,0-120h following chemotherapy
Complete Protection from Both Vomiting and Moderate-to-Severe nausea | 0-24h,24-120h,0-120h following chemotherapy
Time to First Emetic Episode | 0-120h following chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Lin, M.D., Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Fujian Provincial Tumor Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - Jiangsu Provincial Tumor Hospital, Nanjing, Jiangsu
  - The Second Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang
  - Beijing Institute on Thoracic Cancer and Tuberculosis, Beijing

REFERENCES:
- [Derived] Tian W, Wang Z, Zhou J, Zhang S, Wang J, Chen Q, Huang C, Pan L, Zhang L, Huang J, Shen H, Lin T. Randomized, double-blind, crossover study of palonosetron compared with granisetron for the prevention of chemotherapy-induced nausea and vomiting in a Chinese population. Med Oncol. 2011 Mar;28(1):71-8. doi: 10.1007/s12032-009-9398-2. Epub 2010 Jan 5. PMID 20049561
- See also: Publication: Randomized, double-blind, crossover study of palonosetron compared with granisetron for the prevention of chemotherapy-induced nausea and vomiting in a Chinese population. Med Oncol. 2010 Jan 5. [Epub ahead of print] — http://www.ncbi.nlm.nih.gov/pubmed/20049561